CLINICAL TRIAL: NCT02199860
Title: A Double-blind (at Each Dose Level), Randomised, Placebo-controlled, Single Rising Dose Study Investigating the Safety, Tolerability and Pharmacokinetics of Two Spray-dried Formulations of BIBN 4096 BS After Inhalation Administration in Healthy Male and Female Volunteers
Brief Title: Single Rising Dose Study Investigating the Safety, Tolerability and Pharmacokinetics of Spray Dried BIBN 4096 BS After Inhalation Administration in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1149.44
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (4):
- SD I - single rising doses (Experimental)
  Interventions: Drug: SD I
- SD II - single rising doses (Experimental)
  Interventions: Drug: SD II
- SD II - single rising doses + Placebo (Experimental)
  Interventions: Drug: SD II; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SD I
  Arms: SD I - single rising doses
Drug: SD II
  Arms: SD II - single rising doses; SD II - single rising doses + Placebo
Drug: Placebo
  Arms: Placebo; SD II - single rising doses + Placebo

SUMMARY:
The purpose of the present study was to obtain information about the safety, tolerability and pharmacokinetics of BIBN 4096 BS after single inhalation administration of rising doses of spray-dried powder in healthy male and female volunteers. According to the original protocol, the primary objective was to investigate the safety and tolerability of single doses of a new spray-dried inhalation formulation of BIBN 4096 BS (SD I). Following implementation of Amendment 2, this objective was extended to the second spray-dried inhalation formulation SD II with and without concomitant administration of lactose

ELIGIBILITY:
Inclusion Criteria:

Subjects could be included in the study if they met the following criteria:

* Healthy male or female volunteers
* Written informed consent in accordance with Good Clinical Practice (GCP) and the local legislation prior to admission to the study
* Age 21 - 50 years
* Body mass index (BMI): 18.5 - 29.9 kg/m2

Exclusion Criteria:

Subjects were not allowed to participate if any of the following applied:

* Any finding of the medical examination (including blood pressure, pulse rate, Respiratory rate, body temperature and ECG) deviating from normal and of clinical relevance
* Raw > 3 cm H2O • s • L-1 or FEV1 <80% of predicted
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system, psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts,
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (within 1 week prior to administration of investigational drug or during the trial)
* Participation in another trial with an investigational drug (within 2 months prior to drug administration or during the trial)
* Smoker (>10 cigarettes/day or >3 cigars/day or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (>60 gram/day)
* Drug abuse
* Blood donation (≥100 mL within 4 weeks prior to administration of investigational drug or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range and of clinical relevance
* For female subjects:

  * Pregnancy
  * Positive pregnancy test
  * No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device
  * Inability to maintain this adequate contraception during the whole study period,
  * Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2003-05; Primary Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 25 days
Assessment of tolerability on a 4-point scale | 8 days after drug administration
Change in lung function measurements airway resistance (Raw) | up to 5 hours after drug administration
Change in lung function measurement specific conductance (SGaw) | up to 5 hours after drug administration
Change in lunf function measurement forced expiratory volume in 1 second (FEV1) | up to 5 hours after drug administration

SECONDARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 48 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administration
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 48 hours after drug administration
λz (Terminal rate constant in plasma) | up to 48 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTih (Mean residence time of the analyte in the body after inhalation) | up to 48 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 48 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 48 hours after drug administration